CLINICAL TRIAL: NCT04219761
Title: National Tunisian Registry of Percutaneous Coronary Intervention
Acronym: NATURE-PCI
Status: Completed | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Tunisian Society of Cardiology and Cardiovascular Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: DAC-009-NATUREPCI
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: ACS - Acute Coronary Syndrome; Angor Pectoris; Myocardial Infarction; Myocardial Ischemia
Keywords: ACS; PCI; MI
MeSH Terms: conditions — Acute Coronary Syndrome; Angina Pectoris; Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The National Tunisian Registry of Percutaneous Coronary Intervention is an observational, prospective and multicenter study aiming to assess coronary intervention strategies in tunisian departments of cardiology. Cardiologists from both sectors (public and private) are participating in the study, with 37 investigational centers. Data will be captured electronically by DACIMA Clinical Suite, according to FDA 21 CFR part 11 (Food and Drug Administration 21 Code of Federal Regulations part 11), HIPAA (Health Insurance Portability and Accountability Act) & ICH (International Conference on Harmonisation) requirements.

ELIGIBILITY:
Inclusion Criteria:

* Tunisian patient needing PCI (Percutaneous Coronary Intervention) at the enrollment period
* Informed and signed consent

Exclusion Criteria:

* Withdrawn consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tunisian patients needing percutaneous coronray intervention
Sampling Method: Non-Probability Sample
Enrollment: 2698 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
MACE endopoint (Major adverse cardiovascular event) | Time-To-Event measure up to 12 months from baseline
  Composite endpoint (MACE: major adverse cardiovascular event) : occurence of cardiovascular death, or non fatal myocardial infraction, or non fatal stroke, or Target Lesion revascularisation, or Target Vessel Revascularisation

SECONDARY OUTCOMES:
Death | Time-To-Event measure up to 12 months from baseline
  Occurence of death incident (cardiovascular and non cardiovascular)
PCI (Percutaneous Coronary Intervention) | Time-To-Event measure up to 12 months from baseline
  PCI (Percutaneous Coronary Intervention) complications: any side effect event occuring per or post cardiac intervention

CONTACTS AND LOCATIONS:
Overall Officials: Leila Abid, MD, Study Chair — Tunisian Society of Cardiology and Cardiovascular Surgery; Rania Hammami, MD, Principal Investigator — Tunisian Society of Cardiology and Cardiovascular Surgery
Locations (1):
- Société Tunisienne de Cardiologie & de Chirurgie Cardiovasculaire, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hammami R, Boudiche S, Rami T, Ben Halima N, Jamel A, Rekik B, Gribaa R, Imtinene BM, Charfeddine S, Ellouze T, Bahloul A, Hedi BS, Langar J, Ben Ahmed H, Ibn Elhadj Z, Hmam M, Ben Abdessalem MA, Maaoui S, Fennira S, Lobna L, Hassine M, Ouanes S, Mohamed Faouzi D, Mallek S, Mahdhaoui A, Meriem D, Jomaa W, Zayed S, Kateb T, Bouchahda N, Azaiez F, Ben Salem H, Marouen M, Noamen A, Abdesselem S, Hichem D, Ibn Hadj Amor H, Abdeljelil F, Amara A, Bejar K, Khaldoun BH, Hamza C, Ben Jamaa M, Fourati S, Elleuch F, Grati Z, Chtourou S, Marouene S, Sahnoun M, Hadrich M, Mohamed Abdelkader M, Bouraoui H, Kamoun K, Hadrich M, Ben Chedli T, Drissa MA, Charfeddine H, Saadaoui N, Achraf G, Ahmed S, Ayari M, Nabil M, Mnif S, Sahnoun M, Kammoun H, Ben Jemaa K, Mostari G, Hamrouni N, Yamen M, Ellouz Y, Smiri Z, Hdiji A, Bassem J, Ayadi W, Zouari A, Abbassi C, Fatma BM, Battikh K, Kharrat E, Gtif I, Sami M, Bezdah L, Kachboura S, Maatouk MF, Kraiem S, Jeridi G, Neffati E, Kammoun S, Ben Ameur Y, Fehri W, Gamra H, Zakhama L, Addad F, Mohamed Sami M, Abid L. Design and Rationale of the National Tunisian Registry of Percutaneous Coronary Intervention: Protocol for a Prospective Multicenter Observational Study. JMIR Res Protoc. 2022 Aug 5;11(8):e24595. doi: 10.2196/24595. PMID 35930353